CLINICAL TRIAL: NCT06111261
Title: Initial Resuscitation With Albumin in Hemorrhagic Shock to Reduce Positive Fluid Balance: A Randomized Controlled Trial (ABSOLUTE Trial)
Brief Title: Initial Resuscitation With Albumin in Hemorrhagic Shock to Reduce Positive Fluid Balance
Acronym: ABSOLUTE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-Young Oh, Clinical associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2209-086-1359
Record Dates: First submitted 2023-01-10; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Bleeding; Massive Hemorrhage; Massive Transfusion Protocol
Keywords: Massive transfusion protocol; Massive transfusion; Albumin
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin-massive transfusion protocol (Experimental): At the initiation of MTP, 200ml of 20% albumin will be infused followed by transfusion of packed RBC:FFP:Platelet concentrate with ratio of 1:1:1.
  Interventions: Drug: Albumin solution
- Conventional-massive transfusion protocol (Active Comparator): At the initiation of MTP, Balanced crystalloid will be infused followed by transfusion of packed RBC:FFP:Platelet concentrate with ratio of 1:1:1. Albumin will be transfused according to the serum albumin level.
  Interventions: Drug: Balanced crystalloid solution

INTERVENTIONS:
Drug: Albumin solution — 200ml of 20% Human Serum Albumin
  Arms: Albumin-massive transfusion protocol
Drug: Balanced crystalloid solution — Balanced crystalloid solution
  Arms: Conventional-massive transfusion protocol

SUMMARY:
This study is designed to evaluate the effect of early albumin transfusion within massive transfusion protocol on fluid balance and reduced requirement of transfusion.

DETAILED DESCRIPTION:
Eligible patients who require massive transfusion will be randomized in a single-blind manner (participant) in a 1:1 ratio to Conventional Massive Transfusion Pro. tocol group (C-MTP) or Albumin Massive Transfusion Protocol group (A-MTP). When MTP is initiated according to the result of randomization, all patients(or a legal guardian) are informed about the study and potential risks and benefits. Study will be continued only in patients who give informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (19 or older)
* Admitted or planned to admit surgical intensive care unit
* Patients with decreased hemoglobin level more than 20% from baseline within 12 hours, Or
* Patients who are suspected bleeding and hemodynamically unstable requiring more than 0.05mcg/kg/min of norepinephrine infusion to maintain mean blood pressure higher than 65mmHg

Exclusion Criteria:

* Contraindicated to albumin product
* patients with risk factors of increased circulatory volume (heart failure, pulmonary edema, end-stage renal disease with oliguria)
* patients with hemolytic anemia
* History of anaphylactic reaction to blood product

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Total fluid balance until physical hemostasis of bleeding is confirmed (ml) | Time from the initiation of massive transfusion protocol to physical hemostasis of bleeding was confirmed, up to 48 hours after initiation of massive transfusion protocol
  Total fluid balance (Total fluid infused - Total output(urine output, bleeding, drainage, or etc.) until physical hemostasis of bleeding is confirmed (e.g. embolization, surgical exploration and ligation of vessel)

SECONDARY OUTCOMES:
Time from the initiation of massive transfusion protocol to reversal of shock (min) | Time from the initiation of massive transfusion protocol to mean blood pressure was maintained higher than 65mmHg without vasopressor (min), up to 48 hours after initiation of massive transfusion protocol
  Total time required to maintain mean blood pressure higher than 65mmHg without vasopressor
Total amount of fluid until physical hemostasis of bleeding is confirmed (ml) | Time from the initiation of massive transfusion protocol to physical hemostasis of bleeding was confirmed, up to 48 hours after initiation of massive transfusion protocol
  Total amount of transfusion and infusion of albumin product and crystalloid.
Total length of ICU and hospital stay (days) | When discharge from ICU or hospital for any cause (days), through study completion, an average of 4 year
  Total length of ICU and hospital stay
In-hospital mortality | When mortality occurred, through study completion, an average of 4 year
  Mortality occurred during hospital stay
7-day mortality | Within 7 days since the initiation of the massive transfusion protocols
  7-day mortality after the initiation of massive transfusion protocol
28-day mortality | Within 28 days since the initiation of the massive transfusion protocols
  28-day mortality after the initiation of massive transfusion protocol
Acute kidney injury within 2 days of massive transfusion | up to 2 days of MTP
  Incidence of Acute kidney injury (KidneyDisease:ImprovingGlobalOutcomes (KDIGO) stage 1 or above) within 2 days of massive transfusion
Major pulmonary complication within 2 days of massive transfusion | up to 2 days of MTP
  Major pulmonary complication(Pneumonia, PaO2/FiO2 ratio<300, pulmonary edema and pleural effusion) within 2 days of massive transfusion
Transfusion-related adverse event | up to 2 days of MTP
  Transfusion-related adverse event (TRALI, TACO, Anaphylaxis)

CONTACTS AND LOCATIONS:
Overall Officials: Seung-young Oh, M.D., Study Chair — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No